CLINICAL TRIAL: NCT06392425
Title: Role of Serum ADAM 17 (A Disintegrin And Metalloprotease 17) and Caspase 3 in Patients With Chronic Kidney Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, samar salah eldin abdelrahman, Assistant lecturer, Assiut University
Other Study IDs: caspase 3 and ADAM 17 in CKD
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Caspase 3

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- - Group (1): stage(1) CKD patient group: Stage 1 of CKD (eGFR of 90 or greater)
  Interventions: Other: caspase 3 and ADAM 17 biomarkers
- -Group (2): stage (2) CKD patient group: Stage 2 of CKD (eGFR between 60 and 89)
  Interventions: Other: caspase 3 and ADAM 17 biomarkers
- -Group (3) :stage(3) CKD patient group: Stage 3 of CKD (eGFR between 30 and 59)
  Interventions: Other: caspase 3 and ADAM 17 biomarkers
- -Group (4) :stage (4) CKD patient group: Stage 4 of CKD (eGFR between 15 and 29)
  Interventions: Other: caspase 3 and ADAM 17 biomarkers
- -Group (5):stage(5) CKD patient group: Stage 5 of CKD (eGFR less than 15)
  Interventions: Other: caspase 3 and ADAM 17 biomarkers
- -Group (6) :control Group: apparently healthy individuals with matched age and sex are included in this study as a control group for comparison
  Interventions: Other: caspase 3 and ADAM 17 biomarkers

INTERVENTIONS:
Other: caspase 3 and ADAM 17 biomarkers — Role of caspase 3 and ADAM 17 biomarkers in chronic kidney disease

SUMMARY:
1. To evaluate clinical utility of Serum ADAM 17 (A disintegrin and metalloprotease 17) and Caspase 3 measurement in chronic kidney disease patients
2. Study relationship of serum ADAM 17 and Caspase 3 to stages of chronic kidney disease
3. Compare serum ADAM 17 and Caspase 3 levels in Diabetic Chronic kidney disease patients and Non Diabetic Chronic kidney disease patients

DETAILED DESCRIPTION:
Kidney diseases represent a global public health problem ,It is estimated that 10-15% of the population is affected by Chronic kidney disease.(1) Chronic kidney disease (CKD) is defined by persistent urine and structural abnormalities or impaired excretory renal function ( an estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73 m2, persisting for three months or more suggestive of a loss of functional nephrons) (2) the most common contributing factors to CKD include genetic abnormalities and ageing, while the most common underlying diseases associated with CKD are diabetes and hypertension However, CKD can be also due to infectious diseases, autoimmune diseases (such as lupus), and medications (3) A disintegrin and metalloproteinase (ADAM) 17, also known as tumour necrosis factor α-converting enzyme (TACE), is a metalloproteinase that releases the ectodomains of most growth factors, cytokines, receptors and enzymes and has been associated with the presence of chronic kidney disease (5) Clinical and experimental studies have shown that ADAM17 is involved in chronic kidney disease (CKD) with a proinflammatory and profibrotic role, suggesting that it could be an important mediator of CKD progression. ADAM17 inhibition attenuates fibrosis and inflammation, suggesting that its inhibition may be a possible new valuable therapeutic tool in fibrotic kidney disease treatment(6) Caspases (cysteine aspartases, cysteine-aspartic proteases) are protease enzymes which play a role in apoptotic pathway. Their name derives from their specific cysteine protease activity . Most cells have caspases in an inactive proenzyme form, which is activated and induces other pro-caspases, thus initiating a protease cascade. This process is able to amplify the apoptotic signaling pathway and to induce rapid cell death, ,Caspase-3 plays a dominant role in apoptosis, involved in the pathogenesis and progression of chronic kidney disease (CKD).(7)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic kidney disease
2. Patients with different contributing factors e.g Diabetis mellitus, Hypertension ,autoimmune diseases.

Exclusion Criteria:

1. Patients with pulmonary oedema or hepatic disease .
2. Patients with known any organ malignancy.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease with different contributing factors e.g Diabetis mellitus , Hypertension,autoimmune diseases.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-26 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate clinical utility of Serum ADAM 17 (A disintegrin and metalloprotease 17) and Caspase 3 measurement in chronic kidney disease patients | baseline
  Study relationship of serum ADAM 17 and Caspase 3 to stages of chronic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: samar salah, Principal Investigator — Assiut University

REFERENCES:
- [Background] Levin A, Tonelli M, Bonventre J, Coresh J, Donner JA, Fogo AB, Fox CS, Gansevoort RT, Heerspink HJL, Jardine M, Kasiske B, Kottgen A, Kretzler M, Levey AS, Luyckx VA, Mehta R, Moe O, Obrador G, Pannu N, Parikh CR, Perkovic V, Pollock C, Stenvinkel P, Tuttle KR, Wheeler DC, Eckardt KU; ISN Global Kidney Health Summit participants. Global kidney health 2017 and beyond: a roadmap for closing gaps in care, research, and policy. Lancet. 2017 Oct 21;390(10105):1888-1917. doi: 10.1016/S0140-6736(17)30788-2. Epub 2017 Apr 20. PMID 28434650
- [Background] Iino Y. [Definition of CKD and classification of CKD stage]. Nihon Rinsho. 2008 Sep;66(9):1645-9. Japanese. PMID 18788389
- [Background] Thomas MC, Cooper ME, Zimmet P. Changing epidemiology of type 2 diabetes mellitus and associated chronic kidney disease. Nat Rev Nephrol. 2016 Feb;12(2):73-81. doi: 10.1038/nrneph.2015.173. Epub 2015 Nov 10. PMID 26553517
- [Background] Gooz M. ADAM-17: the enzyme that does it all. Crit Rev Biochem Mol Biol. 2010 Apr;45(2):146-69. doi: 10.3109/10409231003628015. PMID 20184396
- [Background] Palau V, Riera M, Duran X, Valdivielso JM, Betriu A, Fernandez E, Pascual J, Soler MJ. Circulating ADAMs are associated with renal and cardiovascular outcomes in chronic kidney disease patients. Nephrol Dial Transplant. 2020 Jan 1;35(1):130-138. doi: 10.1093/ndt/gfy240. PMID 30102333
- [Background] Clementi A, Virzi GM, Manani SM, de Cal M, Battaglia GG, Ronco C, Zanella M. Plasma Cell-Free DNA and Caspase-3 Levels in Patients with Chronic Kidney Disease. J Clin Med. 2023 Aug 28;12(17):5616. doi: 10.3390/jcm12175616. PMID 37685683